CLINICAL TRIAL: NCT06827275
Title: Modifying Feeding Protocols for Critically Ill Patients (mNEED) Based on a Predictive Model of Feeding Intolerance in Critically Ill Patients: a Multicentre, Cohorts Randomized, Controlled Trial
Brief Title: mNEED: a Multicentre, Cluster-randomized, Controlled Trial
Acronym: mNEED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: mNEEDstudy2025; 320.6750.2024-25-6 (Other Grant/Funding Number: Wu Jieping Medical Foundation)
Record Dates: First submitted 2025-01-19; First posted 2025-02-14 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-01

CONDITIONS: Feeding; ICU
Keywords: Nutritional support; prognosis; Feeding intolerance; Intensive care unit; Enteral nutrition

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mNEED (Experimental): mNEED special feeding procedures set by the experimental group
  Interventions: Procedure: Feeding process
- guideline (Active Comparator): Feeding according to the current 2023 ESPEN guidelines
  Interventions: Procedure: Feeding process

INTERVENTIONS:
Procedure: Feeding process — Nutritional therapy is administered according to the feeding procedure

SUMMARY:
Project Name: Improved Feeding Regimen for Critically Ill Patients (mNEED) Based on Feeding Intolerance Prediction Model Solution version number and version date: Version 5.0; 2024.12.16 Informed consent version number and version date: Version 1.0; 2023.10.19

Dear Patient, Recently, the department participated in a nationwide study to develop nutrition protocols for critically ill patients. Participation in a "Modified Feeding Regimen for Critically Ill Patients Based on a Predictive Model of Feeding Intolerance in Critically Ill Patients (mNEED): a multicenter, cohort randomized, controlled trial" is being invited. Before deciding whether to participate in the study, it is important to read the following information carefully to understand the clinical treatment study, its purpose, procedures, duration, and potential benefits, discomforts, and risks. If desired, the information can be discussed with relatives, friends, or the attending physician to assist in making an informed decision. For any questions, please direct them to the physician in charge of the study.

I. Introduction of Clinical Trials

Research Background and Purpose Leading international evidence-based guidelines consistently recommend early targeted nutritional therapy for critically ill patients. However, multicenter cluster-randomized controlled trials (cRCTs) evaluating the impact of implementing these guidelines have not demonstrated patient benefit. In 2022, Ke et al. proposed evidence-based Feeding Guidelines for Critically Ill Patients (NEED), which provided a specific feeding regimen for nutritional therapy in critically ill patients. The results suggested that the NEED group initiated enteral nutrition (EN) earlier and reduced the use of overall parenteral nutrition (PN). However, the NEED feeding strategies did not reduce the incidence of feeding intolerance in critically ill patients.

In previous studies, a predictive model of feeding intolerance (NOFI) in critically ill patients was constructed, demonstrating good predictive power. Therefore, the NEED feeding program will be improved (mNEED) based on NOFI to reduce the occurrence of feeding intolerance (FI) while ensuring the nutritional needs of critically ill patients are met.

Research Process

Research Funds: All treatment methods involved in this study follow conventional treatment procedures, without additional interventions or charges.

Study Content: This study is conducted by the Department of Intensive Care Medicine of the First Hospital of Jilin University, with 2,250 patients expected to be enrolled from ICUs in 90 hospitals nationwide. This study is a multicenter cluster randomized controlled trial, where each center is randomly divided into an experimental group and a control group. Data will be summarized and analyzed statistically.

Possible Risks This study involves an improvement in the feeding strategy for critically ill patients and will not cause additional risks. In the event of serious gastrointestinal adverse events, symptomatic management will be provided promptly.

Subject Benefits All participants in the study will be examined and treated by clinically experienced physicians, who will address questions and provide timely and thoughtful medical services. Participation may lead to improved conditions, and the results of this study may benefit other patients with similar conditions.

Voluntary Participation and Withdrawal Before the trial, a detailed understanding of the clinical trial is encouraged. The hospital and the attending physician are obligated to provide information related to the clinical trial and address any concerns. Participation in the clinical trial treatment is voluntary.

Duty of Confidentiality Medical records (including medical history, physical examination reports, and laboratory results) will be securely stored in the hospital. Access to these records will be limited to physicians (researchers), professional academic committees, ethics committees, and health supervision and management departments. Any public reporting of the study results will not disclose personal identities. Every effort will be made to protect the privacy of personal medical information to the extent permitted by law.

ELIGIBILITY:
Inclusion Criteria:

Age 18 or older Failure of one or more organ systems within 24 hours of admission to the ICU (SOFA score ≥2) Expected to stay in ICU for more than 48 hours Inability to eat orally No EN taboo

ICU Selection Criteria:

ICU in Grade 2 or above hospitals ICU with the ability to carry out intensive care and monitor patient FI ICU type: emergency, medical, surgical, neurosurgical, or comprehensive ICU

Exclusion Criteria:

Patients who have received EN treatment in the past three days AGI Level IV patients Receiving palliative care and expected to die within 48 hours Pregnancy Long-term use of steroids or other immunosuppressants Patients undergoing radiotherapy or chemotherapy for malignant diseases Participation in other clinical studies

ICU Exclusion Criteria:

ICU that refuses to participate in the study ICU that has not passed the ethical review Pediatric ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2250 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Feeding intolerance | Within 7 days in the ICU
  Intolerance to enteral feeding for any clinical reason (vomiting, high gastric residue, diarrhea, gastrointestinal bleeding, etc.). FI should be considered present if at least 20 kcal/kg BW/day via enteral route cannot be reached within 72 h of feeding attempt or if enteral feeding has to be stopped for whatever clinical reason.
  Vomiting: Any visible regurgitation of gastric contents, regardless of volume.
  High Gastric Residual Volume (GRV): GRV > 200 mL per single measurement, assessed every 4 hours via syringe aspiration from the gastric/jejunal tube.
  Diarrhea: Three or more loose or liquid stools per day, with a stool weight greater than 200-250 g/day (or greater than 250 mL/day).
  Gastrointestinal Bleeding: Any bleeding within the gastrointestinal lumen, confirmed by visible blood in vomitus, gastric aspirate, or stool.

SECONDARY OUTCOMES:
Nutrition goal achievement | ICU day 7
  Proportion of Participants Achieving Nutritional Goals (Caloric Intake: 25 kcal/kg/day; Protein Intake: 1.3 g/kg/day) at Day 7 in the ICU Definition: The proportion of critically ill patients achieving at least 80% of their nutritional goals (caloric intake: 25 kcal/kg/day; protein intake: 1.3 g/kg/day) by Day 7 in the ICU. Nutritional intake will be calculated based on daily enteral and parenteral nutrition records, including calorie and protein intake data extracted from electronic medical records or nutrition monitoring tools.
28-day mortality rate | Day 28 after ICU admission
  Death on the 28th day after ICU admission
90-day mortality | Day 90 after ICU admission
  Death on the 90th day after ICU admission
SF-36 (Short Form-36 Health Survey) | Day 28 and 90 after ICU admission
  SF-36 (Short Form-36 Health Survey) Score at Day 28 and Day 90 After ICU Admission Definition: The SF-36 is a widely used, patient-reported survey of health-related quality of life. It consists of 36 items covering eight health domains: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. Each domain is scored on a scale of 0 to 100, with higher scores indicating better health status. The SF-36 score will be assessed at Day 28 and Day 90 after ICU admission.
EuroQol 5 Dimensions 5 Levels (EQ-5D-5L) | Day 28 and 90 after ICU admission
  EuroQol 5-Dimension 5-Level (EQ-5D-5L) Score at Day 28 and Day 90 After ICU Admission Definition: The EQ-5D-5L is a standardized instrument for measuring health-related quality of life. It consists of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels of severity (no problems, slight problems, moderate problems, severe problems, and extreme problems).
diaphragm thickness | ICU day 7
  Measure the thickest part of the diaphragm during inspiration (when inhaling). Use a 5-15 MHz linear array probe positioned between the mid-axillary and anterior axillary lines at the 8th to 11th intercostal spaces, with the marker pointing cephalad. The diaphragm is typically located at a depth of 2 to 4 cm and appears as a three-layered structure between the pleural and peritoneal lines. It is recommended to measure the diaphragm thickness perpendicular to the fibrous direction between the pleural and peritoneal lines, excluding the membrane.
quadriceps thickness | ICU day 7
  With the lower limb lying flat, the midpoint of the line connecting the upper edge of the patella and the anterior superior iliac spine is used as the measurement point. A 5-15 MHz linear array probe is placed perpendicular to the femur, applying minimal probe pressure to avoid deformation of subcutaneous fat and muscle.
rectus femoris cross-sectional area | ICU day 7
  With the lower limb lying flat, the measurement point is located at the lower third of the line connecting the anterior superior iliac spine and the upper edge of the patella. A 5-15 MHz linear array probe is placed perpendicular to the femur, applying minimal probe pressure to avoid deformation of subcutaneous fat and muscle. For patients with a larger muscle cross-sectional area, if the width of the linear probe cannot provide a complete view of the muscle, a convex array probe may be used instead.
upper limb muscle thickness | ICU day 7
  With the upper limb lying flat, the measurement point is located at the lower two-thirds of the distance between the acromion and the antecubital fossa. The thickness measurement includes the biceps brachii and brachialis muscles, spanning from the superficial fascia of the biceps brachii to the uppermost part of the humerus. A 5-15 MHz linear array probe is placed perpendicular to the humerus, applying minimal probe pressure to avoid deformation of subcutaneous fat and muscle.
New infection in ICU | From 48 hours after ICU admission to ICU discharge, assessed up to 90 days
  Incidence of New Infections in the ICU After 48 Hours of Admission Definition: The occurrence of new infections in the ICU, diagnosed after 48 hours of ICU admission, as confirmed by clinical, laboratory, or imaging criteria. Infections include but are not limited to ventilator-associated pneumonia (VAP), catheter-related bloodstream infections (CRBSI), and urinary tract infections (UTI). The observation period will be from 48 hours after ICU admission to ICU discharge, with a maximum assessment period of 90 days.
Length of ICU stay | ICU stay
  Length of ICU Stay Definition: The duration of stay in the ICU, measured in days, from the date of ICU admission to the date of ICU discharge. The maximum observation period will be 90 days.
ventilator-free days | ICU day 28
  The number of days in the ICU during which no ventilator was used

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Hospital of Jilin University, Changchun, Jilin
  - Jilin University, Chaoyang District, Changchun City, Jilin Province, Changchun, Jilin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Y, Li Y, Chen Y, Zhang Y, Feng X, Lv D, Chen Y, Bi X, Yu Y, Peng Y, Li H, Zhang D. Modifying feeding protocols in critically ill patients based on a predictive model of feeding intolerance: protocol for a multicenter cluster randomized controlled trial (the mNEED study). Front Med (Lausanne). 2025 Nov 6;12:1649983. doi: 10.3389/fmed.2025.1649983. eCollection 2025. PMID 41281994